CLINICAL TRIAL: NCT04770792
Title: The Use of 2% Chlorhexidine Gluconate With Mineral Trioxide Aggregate in Indirect Pulp Treatment of Primary Molars: A Randomized Controlled Clinical Trial
Brief Title: The Use of 2% Chlorhexidine Gluconate With Mineral Trioxide Aggregate in Indirect Pulp Treatment of Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Afnan Saber, Principle investigator, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASaber
Record Dates: First submitted 2021-02-09; First posted 2021-02-25 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Indirect Pulp Treatment
Keywords: Indirect pulp treatment; Deep caries; Primary molars; Mineral trioxide aggregate; 2% chlorhexidine gluconate
MeSH Terms: interventions — chlorhexidine gluconate; mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): 2% chlorhexidine gluconate with mineral trioxide aggregate.
  Interventions: Other: 2% chlorhexidine gluconate with mineral trioxide aggregate.
- Control group (Active Comparator): Mineral trioxide aggregate.
  Interventions: Other: Mineral trioxide aggregate.

INTERVENTIONS:
Other: 2% chlorhexidine gluconate with mineral trioxide aggregate. — 2% chlorhexidine gluconate with mineral trioxide aggregate.
  Arms: Experimental group
Other: Mineral trioxide aggregate. — Mineral trioxide aggregate.
  Arms: Control group

SUMMARY:
The aim of this study was to compare the clinical and radiographic success rates of indirect pulp treatment (IPT) performed by combining 2% chlorhexidine gluconate with mineral trioxide aggregate (MTA) versus IPT performed with MTA in children's vital primary molars. A randomized, split-mouth design including 40 children aged 4-8 years was implemented. The study sample composed of 80 primary molars with deep carious lesions. Each child had 1 pair, one tooth from each pair was allocated randomly either to the 2% chlorhexidine gluconate/MTA group or the MTA group. All teeth were restored with stainless steel crowns. Follow-up is carried out to evaluate the teeth clinically and radiographically.

DETAILED DESCRIPTION:
A double blinded, randomized, controlled clinical trial was performed in a split-mouth design. Eighty primary molars in forty subjects were randomly allocated that each subject had one tooth treated with 2% chlorhexidine gluconate and MTA (experimental group), and the other tooth treated with only MTA (control group).

The study was held at King Abdulaziz University Dental Hospital (KAUDH), Jeddah. Forty healthy children with the age range 4- to 8-year-old were included. Each patient had at least two first primary molars or two second primary molars with deep occlusal or proximal caries not approaching the pulp indicated for IPT.

Preoperative periapical radiographs of the teeth considered for treatment in the study were made using extension cone paralleling technique in the x ray machine.

The procedure was performed in two visits by one operator to allow for the setting of MTA. Stainless steel crowns were used as final restorations.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria:

* 4-8 years old.
* Healthy.
* Cooperative.
* Had at least two first primary molars or two second primary molars with deep occlusal or proximal caries not approaching the pulp indicated for IPT.

Teeth inclusion criteria:

* No spontaneous pain.
* No pain on palpation or percussion.
* No signs of fistula or abscess.
* No abnormal mobility.
* No radiolucency at the periapical or interradicular areas.
* No loss of lamina dura.
* No radiographic signs of internal resorption.
* Sufficient tooth structure allowing placement of rubber dam.
* Not expected to exfoliate within 1 year.

Exclusion Criteria:

* Spontaneous pain.
* Pain on palpation or percussion.
* Signs of fistula or abscess.
* Presence of abnormal mobility.
* Radiolucency at the periapical or interradicular areas.
* Loss of lamina dura.
* Radiographic signs of internal resorption.
* No sufficient tooth structure allowing placement of rubber dam.
* Expected to exfoliate within 1 year.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Data Recording Sheet for Intraoral Clinical Examination | 12 months
  Data sheet for recording the clinical outcome criteria obtained by intraoral clinical examination is filled by the investigators. The data sheet includes information regarding the presence or absence of the following:
  1. Spontaneous pain.
  2. Pain on percussion.
  3. Signs of abscess or fistula.
  4. Abnormal mobility. The response for each point is interpreted in the form by either "yes" or "no".
Data Recording Sheet for Periapical Radiographic Evaluation | 12 months
  Data sheet for recording the radiographic outcome criteria obtained from periapical radiograph is filled by the investigators. The data sheet includes information regarding the presence or absence of the following:
  1. Radiolucency at the periapical or interradicular areas.
  2. Loss of lamina dura.
  3. Signs of internal root resorption.
  4. Signs of external pathologic root resorption.
  5. Normal root resorption accompanying the exfoliation process. The response for each point is interpreted in the form by either "yes" or "no".

CONTACTS AND LOCATIONS:
Overall Officials: Afnan M Saber, MSc, Principal Investigator — Phd student at Pediatric Dentistry Department, Faculty of Dentistry, King Abdulaziz University.
Locations (1):
- King Abdulaziz University, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No